CLINICAL TRIAL: NCT01778166
Title: Immuno-enhanced Versus Standard Early Enteral Nutrition Use in Gastrointestinal Postoperative Patients
Brief Title: Gastrointestinal Postoperative Early Enteral Nutrition: Immuno-enhanced Versus Standard Early Enteral Nutrition
Acronym: ISEEN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Danhua Yao, Senior Resident, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ISEEN001; ISEEN (Registry Identifier: ISEEN)
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Gastrointestinal Malignant
Keywords: Early enteral nutrition; Laparoscopic gastrointestinal surgery; Immuno-enhanced nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard early enteral nutrition (Active Comparator): There would be 100 patients in this group
  Interventions: Drug: Standard early enteral nutrition
- Immuno-enhanced early enteral nutrition (Experimental): There would 100 patients in this group
  Interventions: Drug: Immuno-enhanced

INTERVENTIONS:
Drug: Immuno-enhanced — Immediately drip 37°C saline 20 ml/h and exchange to drip 37°C enteral nutrition fluid concerning omega-3-unsaturated fatty acids 20 ml/h at postoperative 6 h via jejunostomy tube or nasogastric tube
  Arms: Immuno-enhanced early enteral nutrition
Drug: Standard early enteral nutrition — Immediately drip 37°C saline 20 ml/h and exchange to drip 37°C standard enteral nutrition fluid 20 ml/h at postoperative 6 h via jejunostomy tube or nasogastric tube
  Arms: Standard early enteral nutrition

SUMMARY:
Patients with gastrointestinal(GI) malignancy usually suffer from malnutrition and suppressed immune function, which might be worsened by major elective surgery.Enteral nutrition has been emphasized for patients with GI malignancy during the perioperative period to accelerate bowel function recovery, and improve nitrogen balance and immune response while reducing postoperative complications and hospitalization time.Early enteral nutrition(EEN) can promote the postoperative recovery of GI function and has been considered to have other advantages such as the reduction of medical cost and maintenance of intestinal barrier function. Immunonutrition containing special compounds like omega-3-unsaturated fatty acids has been put forward to modulate the immune response and improve the immune function in patients with cancer, which may have an better effect on the immune system than standard enteral nutrition. However, studies on immuno-enhanced early enteral nutrition after a resectable GI malignancy surgery are scarce.

The aim of this study was to determine whether immuno-enhanced early enteral nutrition(IEEN) is more effective than standard early enteral nutrition(SEEN) on nutritional status, immune function, surgical outcomes,time to adjuvant chemotherapy and days of hospitalization after laparoscopic GI surgery.

ELIGIBILITY:
Inclusion Criteria:

* Resectable gastric cancer by laparoscope
* Resectable colorectal cancer laparoscope
* Resectable gastrointestinal interstitialoma by laparoscope

Exclusion Criteria:

* Locally unresectable tumor
* Metastatic tumor
* Preoperative total parenteral or enteral nutrition
* Lack of the patient's consent for the trial participation
* Previous gastrointestinal resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Time to tolerate IEEN/SEEN | 30 days after operation

SECONDARY OUTCOMES:
Overall morbidity rate of IEEN/SEEN | 60 days after operation
Mortality rate of IEEN/SEEN after operation | 60 days after operation
Energy metabolism | 10 days after operation
Time to the first postoperative adjuvant chemotherapy | 30 days after operation
Nutritional status in postoperative day1and 7 of IEEN/SEEN | 7 days after operation
Immune function in postoperative day 1 and 7 | 7 days after operation
Postoperative hospital stay length | 60 days after operation
Rehospitalization rate | 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Danhua Yao, MD/PhD, Principal Investigator — Nanjing University
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Osland E, Yunus RM, Khan S, Memon MA. Early versus traditional postoperative feeding in patients undergoing resectional gastrointestinal surgery: a meta-analysis. JPEN J Parenter Enteral Nutr. 2011 Jul;35(4):473-87. doi: 10.1177/0148607110385698. Epub 2011 May 31. PMID 21628607
- [Background] Liu H, Ling W, Shen ZY, Jin X, Cao H. Clinical application of immune-enhanced enteral nutrition in patients with advanced gastric cancer after total gastrectomy. J Dig Dis. 2012 Aug;13(8):401-6. doi: 10.1111/j.1751-2980.2012.00596.x. PMID 22788925
- [Background] Felekis D, Eleftheriadou A, Papadakos G, Bosinakou I, Ferekidou E, Kandiloros D, Katsaragakis S, Charalabopoulos K, Manolopoulos L. Effect of perioperative immuno-enhanced enteral nutrition on inflammatory response, nutritional status, and outcomes in head and neck cancer patients undergoing major surgery. Nutr Cancer. 2010;62(8):1105-12. doi: 10.1080/01635581.2010.494336. PMID 21058198